CLINICAL TRIAL: NCT07293416
Title: Comparative Effects of Neuropilates and Otago Exercises on Balance, Posture and Functional Independence in Individuals With Chronic Stroke
Brief Title: Neuropilates and Otago Exercises on Balance, Posture and Functional Independence in Chronic Stroke
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/S24C14G37016 Zobia Tariq
Record Dates: First submitted 2025-12-08; First posted 2025-12-19 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Chronic Stroke Patients
Keywords: Balance, Chronic Stroke, Functional Independence, Neuropilates, Otago exercises.

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A : Neuropilates (Experimental): This group will receive 50 minutes session of Neuropilates thrice a week for total of eight weeks which will include activation warm-up exercises for 10 minutes, main exercises for 30 minutes and cool-down exercises for 10 minutes
  Interventions: Other: neuropilates
- Group B : Otago Exercise Program (Active Comparator): This group will receive 50 minutes each session of Otago exercise thrice a week for total of eight weeks which will include, muscle strengthening, balance training and 2x week 30 minutes walking session. Depending on the individual's strength and mobility, the exercises will be progressed, by increasing the amount of repetitions or weight
  Interventions: Other: otago exercises

INTERVENTIONS:
Other: neuropilates — 50 minutes session of Neuropilates thrice a week for total of eight weeks which will include activation warm-up exercises for 10 minutes, main exercises for 30 minutes and cool-down exercises for 10 minutes
  Arms: Group A : Neuropilates
Other: otago exercises — 50 minutes each session of Otago exercise thrice a week for total of eight weeks which will include, muscle strengthening, balance training and 2x week 30 minutes walking session. Depending on the individual's strength and mobility, the exercises will be progressed, by increasing the amount of repetitions or weight
  Arms: Group B : Otago Exercise Program

SUMMARY:
This randomized clinical trial will be conducted at various physical therapy clinics of Faisalabad over a six-month period, enrolling a total of 32 participants selected through non probability convenience sampling technique. Participants will be randomly assigned to one of two groups: those undergoing Neuropilates and those performing Otago exercises, with each group consisting of 16 individuals. Assessments will utilize the TUG (Timed Up and Go) to evaluate balance, the Postural Assessment Scale for Stroke Patients (PASS) for posture, and the Functional Independence Measure (FIM) for functional independence. Pre-intervention assessments will establish baseline measures, followed by evaluations at 4 weeks, and post-intervention to track progress. Data analysis will be conducted using SPSS 26 software, allowing for a comprehensive comparison of the interventions' effectiveness. The findings from this study will contribute valuable insights for clinicians and rehabilitation specialists, enhancing therapeutic strategies to support chronic stroke patients in regaining their independence.

DETAILED DESCRIPTION:
Chronic stroke survivors often face profound challenges that considerably impact their balance, posture, and functional independence. These issues can compromise their ability to perform daily activities, reduce their quality of life, and lead to increased dependency on caregivers. Effective rehabilitation strategies are essential for improving these aspects of recovery. Neuropilates, a novel approach that merges the foundational principles of Pilates with targeted neurological rehabilitation techniques, has shown promise in enhancing physical and cognitive function. By focusing on core strength, flexibility, and body awareness, Neuropilates aims to facilitate motor learning and improve overall stability. This study is designed to compare the effectiveness of Neuropilates with Otago exercises-an evidence-based program specifically designed to enhance strength and balance in older adults-on key rehabilitation outcomes for individuals living with chronic stroke. The Otago program emphasizes lower limb strength and balance training, making it a relevant comparison for assessing improvements in functionality.

The randomized clinical trial will be conducted at various physical therapy clinics of Faisalabad over a six-month period, enrolling a total of 32 participants selected through non probability convenience sampling technique. Participants will be randomly assigned to one of two groups: those undergoing Neuropilates and those performing Otago exercises, with each group consisting of 16 individuals. Assessments will utilize the TUG (Timed Up and Go) to evaluate balance, the Postural Assessment Scale for Stroke Patients (PASS) for posture, and the Functional Independence Measure (FIM) for functional independence. Pre-intervention assessments will establish baseline measures, followed by evaluations at 4 weeks, and post-intervention to track progress. Data analysis will be conducted using SPSS 26 software, allowing for a comprehensive comparison of the interventions' effectiveness. The findings from this study will contribute valuable insights for clinicians and rehabilitation specialists, enhancing therapeutic strategies to support chronic stroke patients in regaining their independence.

ELIGIBILITY:
Inclusion Criteria:

* Age 40-70 years
* Both male and female
* Chronic stroke, 6-18 months post-stroke
* Stroke severity score >6 on NIHSS
* MMSE ≥24

Exclusion Criteria:

* • Symptoms of global or receptive aphasia

  * Other neurological disorders: tumors, anoxia, TBI, neurodegenerative diseases, ataxia.
  * Significant cardiorespiratory conditions
  * Currently receiving other complementary interventions
  * Severe motor impairment preventing safe participation

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-04-12 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
The Postural Assessment Scale for Stroke (PASS) | baseline, 4thweek, 8thweek
  The Postural Assessment Scale for Stroke (PASS) is designed to evaluate postural control after stroke. It consists of 12 four-level items assessing the ability to maintain or change positions in lying, sitting, and standing. Scores range from 0 to 36, with 0-12 indicating poor, 13-24 moderate, and 25-36 good postural control. The PASS has excellent inter-rater reliability (α = 0.88, range 0.64-1) and total score reliability (r = 0.99, p < 0.001). Test-retest reliability in chronic stroke patients is also high (ICC = 0.84-0.97).
The Functional Independence Measure (FIM) | baseline, 4thweek, 8thweek
  The Functional Independence Measure (FIM) is used to assess the functional independence of individuals recovering from illness or disability. It includes 18 items covering self-care, mobility, locomotion, communication, and social cognition. Each item is rated on a 7-point scale (1 = total dependence to 7 = complete independence), giving a total score between 18 and 126. Higher scores indicate greater independence. The FIM demonstrates high inter-rater reliability (ICC = 0.86-0.88).
Timed Up and Go (TUG) | baseline, 4thweek , 8thweek
  The Timed Up and Go (TUG) test is a simple, quick, and reliable tool used to assess mobility, balance, and fall risk in individuals with neurological or musculoskeletal conditions. It measures the time taken to stand up from a chair, walk three meters, turn, return, and sit down. A cut-off time of 12 seconds or more indicates a high risk of falling. The test is suitable for people with stroke, Parkinson's disease, multiple sclerosis, hip fracture, or joint replacement. It requires only a chair, stopwatch, and three-meter mark and allows observation of gait, stability, and use of aids. The test shows a sensitivity and specificity of about 87% for identifying fall risk in the elderly population.

CONTACTS AND LOCATIONS:
Overall Officials: Binash Afzal, Principal Investigator — Riphah International University
Locations (3):
- Pakistan (3):
  - Al-Mahmood Physiotherapy Clinic, Faisalabad
  - Faisal Hospital Faisalabad, Faisalabad
  - Syeda Khatoon e Jannat Trust Hospital, Faisalabad

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cronin E, Broderick P, Clark H, Monaghan K. What are the effects of pilates in the post stroke population? A systematic literature review & meta-analysis of randomised controlled trials. J Bodyw Mov Ther. 2023 Jan;33:223-232. doi: 10.1016/j.jbmt.2022.09.028. Epub 2022 Sep 29. PMID 36775522
- [Background] Chen SC, Lin CH, Su SW, Chang YT, Lai CH. Feasibility and effect of interactive telerehabilitation on balance in individuals with chronic stroke: a pilot study. J Neuroeng Rehabil. 2021 Apr 26;18(1):71. doi: 10.1186/s12984-021-00866-8. PMID 33902646